CLINICAL TRIAL: NCT04275726
Title: A Prospective, Multinational, Multicentre, Open-label, Randomised, Non-inferiority Trial to Compare Safety and Effectiveness of Meril's Myval Transcatheter Heart Valve (THV) Series vs. Contemporary Valves (Edwards's Sapien THV Series and Medtronic's Evolut THV Series) in Patients With Severe Symptomatic Native Aortic Valve Stenosis
Brief Title: LANDMARK Trial: a Randomised Controlled Trial of Myval THV
Acronym: LANDMARK
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Meril Life Sciences Pvt. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MLS/MYV-2/LANDMARK; 2020-000137-40 (EudraCT Number)
Record Dates: First submitted 2020-02-04; First posted 2020-02-19 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-04

CONDITIONS: Aortic Valve Stenosis
Keywords: LANDMARK Trial; Trial to evaluate safety & effectiveness of Myval THV; CE Approved Myval THV Series
MeSH Terms: conditions — Aortic Valve Stenosis

STUDY DESIGN:
Intervention Model Description: The randomisation will be carried out with an allocation ratio of 1:1 between Myval THV Series vs. Contemporary Valves (Sapien THV Series and Evolut THV Series).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Myval THV Series (Experimental): Myval THV Series will include Myval/Myval Inception THVs or any subsequent advanced version commercially available at the study site.
  This treatment arm will be assigned to 384 / 768 subjects enrolled in a study.
  Interventions: Device: Myval THV Series
- Contemporary Valves (Active Comparator): * Sapien THV Series will consist of Sapien 3/Sapien 3 Ultra THVs or any subsequent advanced version commercially available at the study site.
  * Evolut THV Series will include Evolut R/Evolut PRO THVs or any subsequent advanced version commercially available at the study site.
  This treatment arm will be assigned to 384 / 768 subjects enrolled in a study.
  Interventions: Device: Contemporary Valves (Sapien THV Series and Evolut THV Series)
- Myval THV Series XL Nested Registry (Experimental): A non-randomised, nested registry of patients with anatomy of native aortic annulus suitable to be implanted with extra-large size of Myval THV series (30.5mm or 32mm) as per Heart Team assessment/Investigator's discretion is designed. The objective of this registry is to assess the safety and effectiveness of extra-large sizes of Myval THV series. Approximately 100 patients will be recruited from approximately 30 participating centres in LANDMARK Trial
  Interventions: Device: Myval THV Series
- Myval THV Series Lead-in Set (Experimental): The Lead-in Set aims to ensure investigators adhere to protocol requirements related to the Myval THV Series device, including imaging and procedural guidelines. Investigators should be independent before enrolling study subjects, allowing for valuable feedback for initial safety assessments. Each investigator must conduct at least two non-randomized lead-in cases under the guidance of an evaluation committee. Lead-in subjects will only receive the study device, and if implantation fails, standard care will be provided. These subjects will not be included in primary or secondary endpoint analyses but will undergo descriptive analysis. Unique numbers will be assigned to all lead-in subjects, and the committee will evaluate outcomes and site independence for future trial recruitment.
  Interventions: Device: Myval THV Series

INTERVENTIONS:
Device: Myval THV Series — The devices in the study are intended to improve aortic valve function for patients with severe symptomatic native aortic valve stenosis who are eligible for TAVR therapy. Every patient must be deemed treatable with an available size of both the test and contemporary heart valves approved for use and commercially available at the investigational centre where the implant procedure is being performed.
  Other Names: Myval/Myval Inception THVs or any subsequent advanced version commercially available at the study site.
  Arms: Myval THV Series; Myval THV Series Lead-in Set; Myval THV Series XL Nested Registry
Device: Contemporary Valves (Sapien THV Series and Evolut THV Series) — The devices in the study are intended to improve aortic valve function for patients with severe symptomatic native aortic valve stenosis who are eligible for TAVR therapy. Every patient must be deemed treatable with an available size of both the test and contemporary heart valves approved for use and commercially available at the investigational centre where the implant procedure is being performed.
  Other Names: Sapien THV Series (Sapien 3/Sapien 3 Ultra THVs) and Evolut THV Series (Evolut R/Evolut PRO THVs ) or any subsequent advanced version commercially available at the study site.
  Arms: Contemporary Valves

SUMMARY:
The primary objective of this study (LANDMARK) is to compare the safety and effectiveness of the Myval THV Series with Contemporary Valves (Sapien THV Series and Evolut THV Series) in patients with severe symptomatic native aortic valve stenosis.

This study will be done in total 768 subjects (384:384, Myval THV Series vs. Contemporary Valves)

The randomisation will be carried out with an allocation ratio of 1:1 between Myval THV Series vs. Contemporary Valves (Sapien THV Series and Evolut THV Series)

DETAILED DESCRIPTION:
LANDMARK Trial is a prospective, randomised, multinational, multicentric, open-label non-inferiority trial of total 768 subjects (384:384, Myval THV Series vs. Contemporary Valves) with severe symptomatic native aortic valve stenosis via transfemoral approach.

* Device sizes applicable for the Myval THV Series: 20 mm, 21.5 mm, 23 mm, 24.5 mm, 26 mm, 27.5 mm, and 29 mm diameter.
* Device sizes applicable for the Sapien 3 THV Series: 20 mm, 23 mm, 26 mm, and 29 mm diameter.
* Device sizes applicable for the Evolut THV Series: 23 mm, 26 mm, 29 mm, and 34 mm diameter.

A non-randomised nested registry will be conducted to include patients requiring extra-large size of Myval THV series (XL Nested Registry)

- Device sizes applicable for the XL Nested Registry: 30.5 mm and 32 mm.

A non-randomized registry will include patients implanted with the Myval THV Series (Lead-in Set).

- The investigators have to perform a minimum of 2 lead-in cases (non-randomised) under the guidance of the lead-in evaluation committee.

ELIGIBILITY:
Inclusion Criteria:

1. Patient ≥18 years of age.
2. Patient or their legal representative has provided written informed consent as approved by the Institutional Review Board (IRB)/Institutional Ethics Committee (IEC) of the investigational site to participate in the study.
3. As per local Heart Team assessment, patient is eligible for TAVI and the patient is suitable for implantation with all three study devices.

Exclusion Criteria:

1. Patients who are not willing to provide informed consent form, or whose legal heirs object to their participation in the study.
2. Any condition, which in the Investigator's opinion, would preclude safe participation of patient in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 988 (Estimated)
Dates: Start 2020-11-04 (Actual); Primary Completion 2024-03-07 (Actual); Study Completion 2033-12-31 (Estimated)

PRIMARY OUTCOMES:
Primary Combined Safety and Effectiveness Endpoint as defined by the Valve Academic Research Consortium-3 (VARC-3) | 30-day
  It is the composite of following:
  * All-cause mortality
  * All stroke
  * Bleeding (Type 3 and 4)
  * Acute kidney injury (AKI) (Stage 2, 3 and 4)
  * Major vascular complications
  * Moderate or severe prosthetic valve regurgitation
  * Conduction system disturbances resulting in a new PPI

SECONDARY OUTCOMES:
The combined safety and effectiveness endpoint as defined by the Valve Academic Research Consortium-3 (VARC-3) | 1-year
  It is the composite of following:
  * All-cause mortality
  * All stroke
  * Bleeding (Type 3 and 4)
  * AKI (Stage 2, 3 and 4)
  * Major vascular complications
  * Moderate or severe prosthetic valve regurgitation
  * Conduction system disturbances resulting in a new PPI
All-cause mortality | Pre-discharge, 30-day, 6-month, 1-year, 2-year, 3-year, 4 year, 5-year, 7-year, and 10-year
  As per VARC-3 defined criteria
All stroke | Pre-discharge, 30-day, 1-year, 3-year, and 5-year
  As per VARC-3 defined criteria
Acute Kidney Injury (AKI) (Stage 2, 3 and 4) | Pre-discharge, 30-day, and 1-year
  As per VARC-3 defined criteria
Bleeding (Type 3 and 4) | Pre-discharge, 30-day, 1-year, 3-year, and 5-year
  As per VARC-3 defined criteria
Moderate or severe prosthetic valve regurgitation | Pre-discharge, 30-day, 1-year, 3-year, 5-year, 7-year, and 10-year
  As per VARC-3 defined criteria
New permanent pacemaker implantation (As per VARC-3 defined criteria) | Pre-discharge, 30-day, 6-month, 1-year, 2-year, 3-year, 4-year, 5-year, 7-year, and 10-year
  o New PPI rates will be analysed further based on the patient's history of left and/or right bundle branch block.
Conduction disturbances and arrhythmias | Pre-discharge, 30-day, 1-year, 3-year, and 5-year
  As per VARC-3 defined criteria
Device success | Pre-discharge and 30-day
  As per VARC-3 defined criteria
Early safety at 30 days | 30-day
  As per VARC-3 defined criteria
Clinical efficacy at 30 days | After 30 days of index procedure
  As per VARC-3 defined criteria
Valve related long-term clinical efficacy | 5-years, 7 years and 10 years
  As per VARC-3 defined criteria
Vascular and access related complications | Pre-discharge, 30-day, and 1-year
  As per VARC-3 defined criteria
Major vascular complications | Pre-discharge, 30-day, and 1-year
  As per VARC-3 defined criteria
Functional improvement from baseline as measured per | [Time frame: Baseline (pre-procedure), 30-day, 1-year, 3-year, 5-year, 7-year, and 10-year], [Time frame: Baseline (pre-procedure), 30-day and 1-year]
  New York Heart Association (NYHA) functional classification [Time frame: Baseline (pre-procedure), 30-day, 1-year, 3-year, 5-year, 7-year, and 10-year] Six-minute walk test [Time frame: Baseline (pre-procedure), 30-day and 1-year]
Echocardiographic endpoints | Baseline, pre-discharge, 30-day, 1-year, 3-year, 5-year, 7-year, and 10-year
  * Effective orifice area (EOA)
  * Index effective orifice area (iEOA)
  * Mean aortic valve gradient
  * Peak aortic valve gradient
  * Peak aortic velocity
  * Total aortic regurgitation, transvalvular regurgitation (except baseline) and paravalvular regurgitation (except baseline)
  * Left ventricular ejection fraction (LVEF)
  * Valve calcification
  * Cardiac output and cardiac index
Bioprosthetic valve deterioration | Pre-discharge, 30-day, 1-year, 3-year, and 5-year
  As per VARC-3 defined criteria
Patient-prosthesis mismatch | Pre-discharge, 30-day, and 1-year
  Severity patient-prosthesis-mismatch will be based on following
  * For subjects with body mass index (BMI) <30 kg/m2, EOAi: 0.85 - 0.66 cm2 /m2 considered as moderate and ≤0.65 cm2 /m2 considered as severe
  * For subjects with BMI ≥30 kg/m2, EOAi: 0.70 - 0.56 cm2 /m2 considered as moderate and ≤0.55 cm2 /m2 considered as severe
  * BMI = weight(kg)/(height (m))2
Length of index hospital stay | At discharge
  o Number of days from hospital admission to discharge.
Re-hospitalization | 30-day, 1-year, 3-year, and 5-year
  As per VARC-3 defined criteria
Health status as evaluated by Quality of Life questionnaires | Baseline (pre-procedure), 30-day, and 1-year
  o 12-Item Short Form Survey (SF-12)
Valve thrombosis | 30-day, 1-year, 3-year, and 5-year
  o Valve thrombosis as per VARC-2 is any thrombus attached to or near an implanted valve that occludes part of the blood flow path, interferes with valve function, or is sufficiently large to warrant treatment. Note that valve-associated thrombus identified at autopsy in a patient whose cause of death was not valve-related should not be reported as valve thrombosis.
Coronary obstruction requiring intervention | Pre-discharge
  As per VARC-3 defined criteria
Valve malpositioning | Pre-discharge
  As per VARC-3 defined criteria
Conversion to open surgery | Pre-discharge
  As per VARC-3 defined criteria
Unplanned use of mechanical circulatory support (cardiopulmonary bypass (CPB), extracorporeal membrane oxygenation (ECMO), transcatheter pumps or intra-aortic balloon pump (IABP) | Pre-discharge
  As per VARC-3 defined criteria
Implantation of multiple (>1) transcatheter valves during the index hospitalization | Index-procedure
  As per VARC-3 defined criteria
Cardiac structural complications | 30 days, 6 months, 1 year, 2 years, 3 years, 4 years, 5 years
  As per VARC-3 defined criteria
Ventricular septal perforation | Pre-discharge
  o Angiographic or echocardiographic evidence of a new septal perforation during or after the TAVI procedure
New onset of atrial fibrillation or atrial flutter | Pre-discharge, 30-day, 1-year, 3-year, and 5-year
  As per VARC-3 defined criteria
Technical success | Post-procedure
  As per VARC-3 defined criteria
Myocardial Infarction | Pre-discharge, 30-day, 1-year, 3-year, and 5-year
  As per VARC-3 defined criteria
Endocarditis | 30-day, 1-year, 3-year, and 5-year
  As per VARC-3 defined criteria

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Baumbach, MD,FESC,FRCP, Study Chair — Barts Heart Center, London, UK; Patrick W. Serruys, MD,PhD,FACC,FESC, Study Director — National University of Ireland, Galway, Ireland
Locations (54):
- Republican Scientific-Practical Centre "Cardiology", Minsk, Belarus
- Hospital Dante Pazanesse, São Paulo, Brazil
- Croatia (2):
  - Split Clinical Hospital Center, Split
  - University Hospital Dubrava Avenija Gojka Šuška 6, Zagreb
- North Estonia Medical Center, Tallinn, Estonia
- France (5):
  - Hôpital Henri Mondor, Créteil
  - Lille University, Lille
  - Institut Cardiovascular Paris-Sud, Massy
  - Arnault Tzanck Institute, Nice
  - Centre Hospitalier Universitaire De Rennes, Rennes
- Germany (7):
  - Kerckhoff-KlinikForschungs GmbH, Bad Nauheim, Hesse
  - Leipzig Heart Institute GmbH, Leipzig, Saxony
  - University Herzentrum Division of Cardiology and Angiology II,University Heart Center Freiburg, Südring 15, Bad Krozingen
  - Klinikum Braunschweig Freisestre, Braunschweig
  - Technology University Dresden Fetscherstraße 76, Dresden
  - Asklepios Kliniken Hamburg Gmbh Lohmuehlenstrasse 5, Hamburg
  - Klinik für Herz-, Thorax- und herznahe Gefäßchirurgie, Universitätsklinikum Regensburg, Regensburg
- Greece (3):
  - Hippkration Hospital, Athens
  - Hygeia hospital, Marousi
  - Interbalkan European Medical Center, Thessaloniki
- Semmelweis University, Budapest, Hungary
- Italy (7):
  - University of Bologna Policlinico S. Orsola-Malpigh, Bologna
  - Policlinico di Catania, Catania
  - San Donato Hospital, Milan
  - San Raffaele Hospital, Milan
  - Clinical Institute Saint Ambrogio, Milan
  - Mauriliano Hospital Largo Filippo, Tortona
  - University Hospital Città della Salute e della Scienza Turin Bramante, Turin
- Netherlands (7):
  - St Antonius Hospital, Nieuwegein, Dutch
  - Radboud University Nijmegen, Nijmegen, Gelderland
  - Isala Zwolle Hospital, Zwolle, Overijssel
  - Onze lieve vrouwe gasthuis Oosterperk 9, Amsterdam
  - Amphia Ziekenhui Hospital, Breda
  - University Medical Center (UMC), Groningen
  - University Medical Center Utrecht, Utrecht
- Auckland City Hospital 2 Park Road, Grafton, Auckland, New Zealand
- Poland (5):
  - John Paul II Hospital, Krakow, Małopolskie Województwo
  - University of Gdansk, Gdansk, Pomorskie Województwo
  - Medical University of Silesia, Katowice, Prussian
  - Institute of Cardiology, Warsaw
  - Uniwersytecki Szpital Kliniczny (USK) Curie-Skłodowskiej 58, Wroclaw
- Portugal (4):
  - Centro Hospitalar Lisboa Ocidental EPE- Hospital Santa Cruz, Av. Prof. Dr. Reinaldo dos Santos, Carnaxide
  - Centro Hospital Lisboa Central E.P.E. - Santa Marta, Lisbon
  - Hospital de Santa Maria, Av. Prof. Egas Moniz MB, Lisbon
  - Centro Hospitalar de Sao Joao, Porto
- University hospital Banska Bystrica Námestie Ludvíka Svobodu 1, Banská Bystrica, Slovakia
- University Medical Center, Ljubljana, Ljubljana, Slovenia
- Spain (5):
  - Hospital Universitari Son Espases Carretera de Valldemossa, Palma de Mallorca, Balearic Islands
  - Hospital Universitario de Gran Canaria Dr Negrin, Las Palmas, Canary Islands
  - Hospital Universitario Renei Sofia, Córdoba
  - Hospital Clínico San Carlos, Madrid
  - Hospital Cliinico Univertistario de Valladolid, Valladolid
- Sweden (2):
  - Sahlgrenska University Hospital, Gothenburg
  - Uppsala University Hospital, Uppsala

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kawashima H, Soliman O, Wang R, Ono M, Hara H, Gao C, Zeller E, Thakkar A, Tamburino C, Bedogni F, Neumann FJ, Thiele H, Abdel-Wahab M, Morice MC, Webster M, Rosseel L, Mylotte D, Onuma Y, Wijns W, Baumbach A, Serruys PW. Rationale and design of a randomized clinical trial comparing safety and efficacy of myval transcatheter heart valve versus contemporary transcatheter heart valves in patients with severe symptomatic aortic valve stenosis: The LANDMARK trial. Am Heart J. 2021 Feb;232:23-38. doi: 10.1016/j.ahj.2020.11.001. Epub 2020 Nov 6. PMID 33160946
- [Background] Tobe A, Onuma Y, Soliman O, Baumbach A, Serruys PW. LANDMARK trial: Update in study protocol. Am Heart J. 2024 Apr;270:162-163. doi: 10.1016/j.ahj.2024.02.008. Epub 2024 Feb 16. No abstract available. PMID 38369219
- [Result] Baumbach A, van Royen N, Amat-Santos IJ, Hudec M, Bunc M, Ijsselmuiden A, Laanmets P, Unic D, Merkely B, Hermanides RS, Ninios V, Protasiewicz M, Rensing BJWM, Martin PL, Feres F, De Sousa Almeida M, van Belle E, Linke A, Ielasi A, Montorfano M, Webster M, Toutouzas K, Teiger E, Bedogni F, Voskuil M, Pan M, Angeras O, Kim WK, Rothe J, Kristic I, Peral V, Garg S, Elzomor H, Tobe A, Morice MC, Onuma Y, Soliman O, Serruys PW; LANDMARK trial investigators. LANDMARK comparison of early outcomes of newer-generation Myval transcatheter heart valve series with contemporary valves (Sapien and Evolut) in real-world individuals with severe symptomatic native aortic stenosis: a randomised non-inferiority trial. Lancet. 2024 Jun 22;403(10445):2695-2708. doi: 10.1016/S0140-6736(24)00821-3. Epub 2024 May 22. PMID 38795719
- [Result] Royen NV, Amat-Santos IJ, Hudec M, Bunc M, Ijsselmuiden A, Laanmets P, Unic D, Merkely B, Hermanides RS, Ninios V, Protasiewicz M, Rensing BJWM, Martin PL, Feres F, Sousa M, Belle EV, Linke A, Ielasi A, Montorfano M, Webster M, Toutouzas K, Teiger E, Bedogni F, Voskuil M, Pan M, Angeras O, Kim WK, Rothe J, Kristic I, Peral V, Van den Branden BJL, Westermann D, Bellini B, Garcia-Gomez M, Tobe A, Tsai TY, Garg S, Thakkar A, Chandra U, Morice MC, Soliman O, Onuma Y, Serruys PW, Baumbach A. Early outcomes of the novel Myval THV series compared to SAPIEN THV series and Evolut THV series in individuals with severe aortic stenosis. EuroIntervention. 2025 Jan 20;21(2):e105-e118. doi: 10.4244/EIJ-D-24-00951. PMID 39589296
- [Derived] Serruys PW, Tobe A, van Royen N, Amat-Santos IJ, Hudec M, Bunc M, Van den Branden BJL, Laanmets P, Unic D, Merkely B, Hermanides RS, Ninios V, Protasiewicz M, Rensing BJWM, Martin PL, Feres F, De Sousa Almeida M, van Belle E, Linke A, Ielasi A, Montorfano M, Webster M, Toutouzas K, Teiger E, Bedogni F, Voskuil M, Pan M, Angeras O, Kim WK, Rothe J, Abdel-Wahab M, Kristic I, Peral V, Garg S, Tsai TY, Thakkar A, Chandra U, Smits PC, Morice MC, Onuma Y, Baumbach A; LANDMARK Investigators. 1-Year Outcomes of Novel Balloon-Expandable vs Contemporary Transcatheter Heart Valves in Severe Aortic Stenosis: The LANDMARK Trial. J Am Coll Cardiol. 2025 Nov 16:S0735-1097(25)10159-9. doi: 10.1016/j.jacc.2025.10.076. Online ahead of print. PMID 41384893
- [Derived] Soliman O, Hasabo EA, van Royen N, Amat-Santos IJ, Hudec M, Bunc M, IJsselmuiden A, Laanmets P, Unic D, Merkely B, Hermanides RS, Mouden M, Ninios V, Protasiewicz M, Rensing BJWM, Martin PL, Feres F, Almeida MS, van Belle E, Linke A, Ielasi A, Montorfano M, Webster M, Toutouzas K, Teiger E, Bedogni F, Voskuil M, Rubio DM, Angeras O, Kim WK, Rothe J, Kristic I, Peral V, Van den Branden BJL, Thakkar A, Chandra U, Neiroukh D, Ayhan C, Nosir MY, Yacoub MS, Ali S, Altamimi M, Elzomor H, Serruys PW, Baumbach A. Comparative 30-day echocardiographic outcomes of Myval vs. Sapien and Evolut THVs: insights from LANDMARK trial. Eur Heart J Cardiovasc Imaging. 2026 Feb 9;27(2):247-260. doi: 10.1093/ehjci/jeaf245. PMID 40875489
- [Derived] Kawashima H, Wang R, Mylotte D, Jagielak D, De Marco F, Ielasi A, Onuma Y, den Heijer P, Terkelsen CJ, Wijns W, Serruys PW, Soliman O. Quantitative Angiographic Assessment of Aortic Regurgitation after Transcatheter Aortic Valve Implantation among Three Balloon-Expandable Valves. Glob Heart. 2021 Mar 19;16(1):20. doi: 10.5334/gh.959. PMID 33833944
- See also: Rationale and design of a randomized clinical trial comparing safety and efficacy of myval transcatheter heart valve versus contemporary transcatheter heart valves in patients with severe symptomatic aortic valve stenosis: The LANDMARK trial — https://pubmed.ncbi.nlm.nih.gov/33160946/
- See also: LANDMARK comparison of early outcomes of newer-generation Myval transcatheter heart valve series with contemporary valves (Sapien and Evolut) in real-world individuals with severe symptomatic native aortic stenosis:a randomised non-inferiority trial. — https://pubmed.ncbi.nlm.nih.gov/38795719/
- See also: Early outcomes of the novel Myval THV series compared to SAPIEN THV series and Evolut THV series in individuals with severe aortic stenosis. EuroIntervention — https://pubmed.ncbi.nlm.nih.gov/39589296/
- See also: LANDMARK trial: Update in study protocol. — https://pubmed.ncbi.nlm.nih.gov/38369219/